CLINICAL TRIAL: NCT07218224
Title: Expanded Access:18F-Fluorocholine for the Detection of Parathyroid Adenomas
Status: Available | Type: Expanded Access
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: 25-44398
Record Dates: First submitted 2025-10-02; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Parathyroid Adenomas
MeSH Terms: conditions — Parathyroid Neoplasms | interventions — fluorocholine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: 18F-Fluorocholine (FCH) — A dose of 4-7 millicurie (mCi) +/- 10% of radiotracer 18F-Fluorocholine (FCH) manufactured at UCSF will be given intravenously.
  Other Names: FCH; 18F-fluorocholine (fluoromethyl-(2-hydroxyethyl)-dimethylazanium)
Procedure: Positron emission tomography (PET) — A scan is a procedure that produces images of organs and tissues used in conjunction with a radiotracer.
  Other Names: PET Scan

SUMMARY:
This expanded access protocol is proposed to allow University of California San Francisco (UCSF) patients additional access to 18F-fluorocholine (FCH) Positron Emission Tomography (PET) imaging for localization of parathyroid adenomas.

DETAILED DESCRIPTION:
No health outcome measures will be obtained under this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 13 years.
2. Evidence of primary hyperparathyroidism.
3. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco